CLINICAL TRIAL: NCT00262678
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of EN3267 for the Treatment of Breakthrough Pain in Opioid Tolerant Cancer Patients.
Brief Title: Efficacy and Safety of Sublingual Fentanyl Tablets in Treatment of Breakthrough Pain in Cancer Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EN3267-005
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Pain; Cancer
MeSH Terms: conditions — Pain; Neoplasms

INTERVENTIONS:
Drug: EN3267

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of sublingual fentanyl tablets in relieving breakthrough pain in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 17 years of age or older
* Stable cancer-related pain.
* Are receiving a stable, fixed-schedule oral opioid regimen equivalent to 60 to 1000 mg of oral morphine per day or transdermal fentanyl therapy equivalent to 50 to 300 µg/h, and are on a stable dose of opioid medication for relief of breakthrough pain for at least 14 days prior to screening.
* Experiencing 1-4 episodes of breakthrough pain per day.
* Meet the criteria defined in the Eastern Cooperative Oncology Group (ECOG) Performance Status for Grade 0, 1, or 2.

Exclusion Criteria:

* Are pregnant or lactating.
* Have uncontrolled or rapidly escalating pain.
* Have moderate to severe ulcerative mucositis.
* Have a cardiopulmonary disease that would increase the risk of administering potent opioids.
* Have neurologic or psychologic disease that would compromise data collection
* Have any clinically significant condition that would, in the investigator's opinion, preclude study participation.
* Are currently taking monoamine oxidase inhibitors (MAOIs), or have taken MAOIs within 14 days prior to enrolling in the study.
* Have received strontium 89 therapy within 60 days prior to entering the study.
* Have received anti-neoplastic therapy within 2 weeks of study entry that, in the investigator's opinion, will influence assessment of breakthrough pain
* Have received any investigational drug (non-approved) within 30 days prior to the first dose of study medication, or are scheduled to receive an investigational drug other than EN3267 during the course of the study.
* Have hypersensitivities, allergies, or contraindications to fentanyl.
* Have a significant prior history of substance abuse or alcohol abuse.
* May have difficulty complying with the protocol, as assessed by the investigator.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-12; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Carolinas Pain Institute, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Rauck RL, Tark M, Reyes E, Hayes TG, Bartkowiak AJ, Hassman D, Nalamachu S, Derrick R, Howell J. Efficacy and long-term tolerability of sublingual fentanyl orally disintegrating tablet in the treatment of breakthrough cancer pain. Curr Med Res Opin. 2009 Dec;25(12):2877-85. doi: 10.1185/03007990903368310. PMID 19814586